CLINICAL TRIAL: NCT04289740
Title: Transdiagnostic Group Cognitive Behavioral Therapy Versus Group Relaxation Therapy for Adolescents With Emotional Disorders (PsicAP-A): Protocol
Brief Title: Transdiagnostic Group Cognitive Behavioral Therapy (PsicAP-A) for Adolescents With Emotional Disorders
Acronym: PsicAP-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Hospital de laredo (Unknown); Hospital Sierrallana (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PsicAP-A
Record Dates: First submitted 2020-02-11; First posted 2020-02-28 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Emotional Disorder
Keywords: emotional disorders; cognitive behavioural therapy; adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive-bahavioral therapy (Experimental): Trasdiagnotic cognitive-behavioral group therapy: The psychological interventions will be manualized. Patients assigned to the experimental group will receive 7 sessions (1.5 hr/session) in groups of approximately 8-10 individuals over a 12 week period.
  Interventions: Behavioral: 7 sessions (1.5 hr/session) in groups of approximately 8-10 individuals
- relaxation therapy (Active Comparator): The control group will receive a progressive muscle relaxation group intervention, based on the Bernstein and Borkoveck procedure. This intervention will have the same number of sessions as the experimental intervention and last anywhere from 60 to 90 minutes, depending on the session.
  Interventions: Behavioral: a progressive muscle relaxation group intervention, based on the Bernstein and Borkoveck procedure plus same number of sessions as the experimental intervention.

INTERVENTIONS:
Behavioral: 7 sessions (1.5 hr/session) in groups of approximately 8-10 individuals — Patients assigned to the experimental group will receive 7 sessions (1.5 hr/session) in groups of approximately 8-10 individuals over a 12 week period
  Arms: cognitive-bahavioral therapy
Behavioral: a progressive muscle relaxation group intervention, based on the Bernstein and Borkoveck procedure plus same number of sessions as the experimental intervention. — The control group will receive a progressive muscle relaxation group intervention, based on the Bernstein and Borkoveck procedure. This intervention will have the same number of sessions as the experimental intervention and last anywhere from 60 to 90 minutes, depending on the session.
  Arms: relaxation therapy

SUMMARY:
Emotional disorders such as anxiety and depression are highly prevalent during adolescence and associated with functional impairment that commonly extends into adulthood. In the primary care (PC) setting, these disorders are frequently underdiagnosed and undertreated. Objective: To carry out a prospective, randomized controlled trial (RCT) to test the efficacy of a new transdiagnostic cognitive behavioural group therapy (TD-CBT) protocol for adolescents (age 12 to 18 years) compared to group relaxation therapy (RT). Methods: Two-arm, single-blind, RCT (expected N=160) to compare group TD-CBT for emotional disorders to group RT. The group TD-CBT will be administered in seven sessions (90 min/session) over 12 weeks. Psychological assessments will be carried out at baseline, post-treatment, and at months 3, 6, and 12 after treatment. The assessments will include measures of depression, anxiety, somatization, quality of life, disability, and cognitive-emotional factors. The study will be conducted in two PC centres located in Cantabria, Spain. Discussion: This is the first RCT to evaluate the efficacy of group TD-CBT for emotional disorders in adolescents in the PC setting in Spain. If, as expected, the results confirm the superiority of TD-CBT to conventional RT, the widespread implementation of this new approach-based on scientific evidence obtained in a real-world, primary care setting-could improve treatment outcomes and quality of life in adolescents suffering from anxiety or depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 to 17, inclusive, who present to the PC centre seeking treatment for symptoms of anxiety or depression.
* Scores above the predetermined cut-off points on the GAD-7 (>= 5) and PHQ-9 (>= 5).
* Agreement to participate in the study, with written informed consent provided by both patients and parents/guardians.

Exclusion Criteria:

* Presence of any severe mental disorder, including autism spectrum disorders, bipolar disorder, schizophrenia, anorexia nervosa, substance dependence, personality disorder, and major depressive disorder (PHQ-9> 20).
* Presence of severe or recent suicide attempts
* Moderate or severe behaviour disorder that could interfere with the dynamics of the therapy groups.
* Presence of a mental disability (IQ < 75).
* Be receiving psychological treatment or any type of specialized care related to mental health.
* Receiving any psychopharmacological treatment.
* Parents involved in legal litigation due to separation or divorce.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | 12 month follow-up period.
  Patient Health Questionnaire - 9 item (PHQ-9), adolescent version. Nine items assessing depressive symptoms with Likert response with values ranging from 0 to 3 (Total score range: 0-27; higher scores means a worse outcome)
Depressive symptoms | 12 month follow-up period.
  Children's Depression Inventory, short version (CDI-S). Consists of 10 items answered on a three-point scale, where 0 = absence of the symptom, 1 = moderate symptom, and 2 = severe symptom. The total score ranges from 0 to 20. Higher scores means a worse outcome
Anxiety symptoms | 12 month follow-up period.
  Generalized Anxiety Disorder - 7 item (GAD-7). It is composed of 7 Likert response items, ranging from 0 to 3 points (Total score range: 0-21). Higher scores means a worse outcome.
Anxiety symptoms | 12 month follow-up period.
  Spence Children Anxiety Scale, short version (SCAS-S). It consists of 19 items, ranging from 0 to 3, as follows: 0 = "never", 1 = "sometimes", 2 = "many times", 3 =" always". Total scores range from 0-57 points. Higher scores means a worse outcome.

SECONDARY OUTCOMES:
the Quality of life | 12 month follow-up period.
  KIDSCREEN-10 index. It is composed of 10 Likert response items, ranging from 1 to 5 points. (Total score range: 10-50). Higher scores means a better outcome.
Somatizations | 12 month follow-up period.
  PHQ-15. is composed of 15 Likert response items, ranging from 0 to 2 points. (Total score range: 0-30). Higher scores means a worse outcome.
Rumination | 12 month follow-up period.
  Ruminative Responses Scales (RRS), brooding subscale. It is composed of 5 Likert response items, ranging from 1 to 4 points. (Total score range: 5-20). Higher scores means a worse outcome.
Pathological worry | 12 month follow-up period.
  Penn State Worry Questionnaire (PSWQ), reduced 8-item version. It is composed of 8 Likert response items, ranging from 1 to 5 points. (Total score range: 5-40). Higher scores means a worse outcome.
Attentional and interpretative biases | 12 month follow-up period.
  Inventory of Cognitive Activity in Anxiety Disorders (IACTA), abbreviated 5-item version. It is composed of 5 Likert response items, ranging from 0 to 4 points. (Total score range: 0-20). Higher scores means a worse outcome.
Emotional regulation | 12 month follow-up period.
  Emotion Regulation Questionnaire (ERQ). It is composed of 10 Likert response items, ranging from 1 to 7 points. It assess two emotion-regulation strategies: cognitive reappraisal (6 items; range 6-42; higher scores means a better outcome) and expressive suppression (4 items; range 4-28: higher scores means a worse outcome)
Metacognitive beliefs | 12 month follow-up period.
  Metacognitions Questionnaire (MCQ-30); the 6-item negative metacognitive beliefs subscale.
  It is composed of 6 Likert response items, ranging from 1 to 4 points. (Total score range: 6-24). Higher scores means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - centro salud mental Girones, Girona
  - Centro Salud Mental Selva Marítima, Girona
  - Hospital de Laredo, Laredo
  - Hospital Sierrallana, Torrelavega

IPD SHARING:
Plan to Share IPD: No